CLINICAL TRIAL: NCT06218368
Title: A Cluster Randomized Controlled Trial to Evaluate the Effectiveness of an Educational Toolkit Among Poor Communities in Improving Vaccination Confidence in the Philippines
Brief Title: A Tool Kit to Improve Vaccine Confidence in the Philippines
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: International Care Ministries, the Philippines (Unknown)
Responsible Party: Principal Investigator, Xiaolin Wei, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRCT2021710
Record Dates: First submitted 2023-12-17; First posted 2024-01-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Measles; Polio; Vaccination Hesitancy
MeSH Terms: conditions — Measles; Poliomyelitis; Vaccination Hesitancy | interventions — Poliovirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive our vaccine toolkit intervention, which includes two main components: 1) our educational toolkit on MMR and polio vaccination in the form of a video, which will be introduced and presented to the participants from Week 12 to Week 15 of the Transform program, 2) reminding messages regarding vaccination, which will be delivered following the video session and embedded in Saving Groups program run in the communities. Additionally, participants in the intervention arm will also receive a series of 15 soap opera videos, one for each week, to complement the 15-week Transform Program's education session, which is the core intervention of the Soap Opera Trial developed and run by the ICM.
  Interventions: Behavioral: Educational toolkit on MMR and polio vaccination
- Control (No Intervention): In the control group, participants will attend the standard 15-week Transform program, with education sessions delivered through traditional lectures by health educators from ICM on the topics of income creation, education, food security, and resilience. Our educational toolkit of MMR and polio vaccination will not be provided and there will be no specific reminders or discussions regarding MMR and polio vaccinations.

INTERVENTIONS:
Behavioral: Educational toolkit on MMR and polio vaccination — The educational video about vaccines was adapted from a health educational toolkit that aims to promote community confidence in vaccines in the ultra-poor Philippine households. This toolkit contains persuasive messaging on vaccination guidelines, vaccines safety and efficacy, and myths and misconceptions of MMR and polio vaccines. Participants in the intervention arm will receive our educational video about MMR and polio vaccines. Additionally, health educators from ICM will teach the participants to understand their vaccination cards and orally remind them to have their children vaccinated at each week's Transform Program session from week 12 until week 15. After the end of the Transform Program, about 40-50% of the participants in the intervention arm will attend another community-based program run by ICM called the Savings Groups, where the participants will receive weekly reminding messages about MMR and polio vaccination in their group meetings for three months.
  Arms: Intervention

SUMMARY:
This cluster randomized controlled trial (RCT) aims to evaluate the feasibility and efficacy of an educational toolkit in enhancing measles, mumps, rubella (MMR) and polio vaccine confidence in the Philippines. The toolkit contains four aspects: an introduction to MMR and polio vaccines, vaccine safety and efficacy, vaccination guidelines (including schedules and locations), and debunking myths and misconceptions. Presented as a 10-minute video and followed by reminder messages from health educators, the toolkit was developed in collaboration with International Care Ministries (ICM) health educators and translated into local dialects.

Our toolkit will be embedded in a RCT called the Soap Opera Trial, which is designed and run by the ICM leveraging their community-based Transform Program. The standard Transform Program consists of 15 weeks of education sessions delivered by local health educators through traditional lectures in each community. The trial aims to evaluate the impact of a variation to their standard Transform Program, which uses aspirational videos to deliver education about food security, livelihood, and health. The soap opera to be shown in the video includes drama and plot twists similar to a typical television show but highlights lessons about income creation, health care, and resilience, which are key behaviors and outcomes that can help the poor lift themselves out of poverty. The ICM will conduct this RCT to assess the impact of these soap opera videos on outcomes such as aspirations about the future. A total of 180 communities participating in the Transform program will be randomly assigned to one of the two arms. In the intervention arm, the participants will receive our vaccine toolkit intervention (including educational video and reminding messages about MMR and polio vaccines) and 15 soap opera videos alongside standard Transform Program, while participants in the control arm will receive the standard Transform Program, in which the education sessions are delivered through lectures.

The effectiveness of the toolkit will be evaluated by 1) the rate of MMR and polio vaccination among children of the Transform Program participants and 2) knowledge and attitudes towards these vaccines among the participants. Additionally, the relevance, applicability, and feasibility of the toolkit will be assessed using qualitative research methods, and cost-effectiveness of the intervention will be assessed.

DETAILED DESCRIPTION:
This cluster randomized controlled trial (RCT) aims to assess the feasibility and efficacy of an educational toolkit co-developed with local stakeholders to enhance confidence in measles, mumps, rubella (MMR) and polio vaccines in the Philippines. The toolkit contains information and messages about the following four aspects of MMR and polio vaccines: 1) comprehensive introduction of MMR and polio; 2) vaccines safety and efficacy; 3) MMR and polio vaccination guidelines with vaccination schedules and locations; and 4) myths and misconceptions. The educational toolkit will be presented using a 10-minute translated video converted from PowerPoint slides in one session. Reminder messages regarding vaccination will then be delivered in following sessions by health educators. The educational toolkit, as well as the adapted PowerPoint slide deck and accompanying script, was collaboratively developed with health educators from International Care Ministries (ICM). Professional translators have translated the finalized English version of the slide deck and script into the local dialects. Subsequently, ICM produced a video featuring a health worker presenting the toolkit, synchronized with the voiceover and PowerPoint slides.

Our toolkit will be embedded in a RCT called the Soap Opera Trial, which is designed and run by the ICM leveraging their community-based Transform Program. The standard Transform Program consists of 15 weeks of education sessions delivered by local health educators through traditional lectures in each community. The trial aims to evaluate the impact of a variation to their standard Transform Program, which uses aspirational videos to deliver education about food security, livelihood, and health. The soap opera to be shown in the video is entitled "First Light" and is produced by ICM's own internal media team. It includes drama and plot twists similar to a typical television show but highlights lessons about income creation, health care, and resilience, which are key behaviors and outcomes that can help the poor lift themselves out of poverty. The ICM will conduct this cluster RCT to assess the impact of these soap opera videos on outcomes such as aspirations about the future, investments on children's education, social capital, health, hope, and economic outcomes. A 'cluster' is defined as a community participating in the Transform Program. Each community consists of 30 participants, forming the basic unit for our intervention and analysis. Randomization will be performed at the community level by the ICM, and the 180 communities participating in the Transform program will be randomly assigned to one of the two arms (intervention and control). In the intervention arm, the participants will receive our vaccine toolkit intervention (including educational video and reminding messages about MMR and polio vaccines) and 15 soap opera videos alongside standard Transform Program, while participants in the control arm will receive the standard Transform Program, in which the education sessions are delivered through lectures.

The effectiveness of the toolkit will be evaluated by 1) the rate of measles, mumps, rubella (MMR) and polio vaccination among children of the Transform Program participants and 2) knowledge and attitudes towards these vaccines among the participants. Differences in the two outcomes will be compared between the intervention and control arms using appropriate statistical analysis. Additionally, the relevance, applicability, and feasibility of the toolkit will be assessed using qualitative research methods. The investigators will purposively select 30 end-users to conduct semi-structured interviews, which aim to understand the accuracy and appropriateness of the toolkit content, user perception of the toolkit's relevance, and overall satisfaction with the toolkit. Finally, the investigators will conduct a cost-effectiveness analysis to compare the cost, participants' attitude towards MMR and polio vaccines, and the immunization rates of children in the immediate families of participants associated with our intervention versus no intervention over the entire intervention time horizon.

ELIGIBILITY:
Inclusion criteria

* Individuals reside in the participating communities where ICM recruits for the Transform Program.
* Individuals meet the criteria and definition of ultra-poor based on the ICM's screening*.
* Individuals give oral informed consent to participate in the health education sessions which includes the delivery of our toolkit. There must be 30 eligible participants before a community will be approved to participate in the ICM Transform Program.

  * All participating communities of the ICM Soap Opera trial who provided consents to health education sessions will be eligible to participate in the vaccine confidence trial. Participants will be screened using a poverty score card, loosely based on the Progress out of Poverty Index (PPI) developed for the Philippines (Innovations for Poverty Action, 2014) and self-reported household income. Participants in households that meet the definition of ultra-poor by income (< 22 Philippine pesos per person per day) are prioritized to be recruited for the Transform Program.

Exclusion criteria:

- Individuals who refuse to participate will not be included in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5400 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
First-dose measles-containing-vaccine (MCV) coverage rate | 6 months after intervention
  The rate of first-dose measles-containing-vaccine (MCV) vaccination among children aged 12 months among the family of participants

SECONDARY OUTCOMES:
Two-dose MCV coverage rate | 6 months after intervention
  Two-dose MCV coverage rate among participants' children over 24-month old
Polio vaccination rate | 6 months after intervention
  The rate of polio vaccination among children over 14 weeks old who have received at least three doses of polio vaccines (IPV or OPV) among the family of participants
Mean knowledge score | 6 months after intervention
  Mean knowledge score towards measles and polio vaccines among the participants, measured by a 10-item questionnaire developed by the investigators

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Wei, PhD, Principal Investigator — University of Toronto
Locations (1):
- International Care Ministries, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Yes
According to the ethical agreements, the data is only available for research purpose of the study team. Individual patient data cannot be posted and downloaded in a public data depository. Anonymous data can be shared upon request to the study contacts with joint ethics application to the University of Toronto.
Supporting Information: Study Protocol, SAP
Time Frame: After publication in peer-reviewed journals.
Access Criteria: The research team will aim to publish them in open access journals as priority so that all other researchers will freely access to them.

REFERENCES:
- [Derived] Wu S, Dong Q, Zhang Z, Pang S, Thorpe K, Kelly M, Haldane V, Lau L, Wei X. Effectiveness of an Education Toolkit Delivered by Soap Operas Among Communities Living in Extreme Poverty in Improving Vaccination Confidence in the Philippines: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 30;14:e77022. doi: 10.2196/77022. PMID 41166704